CLINICAL TRIAL: NCT00070538
Title: A Phase I Study Of VNP40101M And Cytarabine For Patients With Hematologic Malignancies
Brief Title: VNP40101M and Cytarabine in Treating Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: VION-CLI-034; CDR0000334879 (Registry Identifier: PDQ (Physician Data Query)); MDA-2003-0326
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2008-08

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: recurrent adult acute lymphoblastic leukemia; blastic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; chronic myelomonocytic leukemia; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; untreated adult acute lymphoblastic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — Cytarabine; laromustine

INTERVENTIONS:
Drug: cytarabine
Drug: laromustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as VNP40101M and cytarabine, use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of combining VNP40101M with cytarabine in treating patients who have hematologic malignancies, including myelodysplastic syndrome or relapsed, refractory, or untreated leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of VP40101M when administered with cytarabine in patients with hematologic malignancies.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is an open-label, dose-escalation study of VNP40101M.

Patients receive cytarabine IV over 24 hours on days 1-4 for patients under 65 years of age OR on days 1-3 for patients 65 years of age and over. Patients also receive VNP40101M IV over 15-60 minutes on day 2. Treatment repeats every 4 weeks for up to 3 courses (in patients with responding disease) in the absence of disease progression or unacceptable toxicity. Patients with a continued response may receive additional courses at the discretion of the investigator.

Cohorts of 3-6 patients receive escalating doses of VNP40101M until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 10 patients may receive treatment at the MTD.

PROJECTED ACCRUAL: Approximately 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of leukemia or myelodysplastic syndromes (MDS) meeting criteria for 1 of the following:

  * Relapsed or refractory leukemia for which there is no standard therapy anticipated to result in a durable remission

    * Acute myeloid leukemia
    * Acute lymphocytic leukemia
    * Chronic myelogenous leukemia

      * In blast crisis
  * Untreated leukemia and standard therapy is refused
  * Any of the following poor-risk MDS:

    * Refractory anemia with excess blasts (RAEB)
    * RAEB in transformation
    * Chronic myelomonocytic leukemia
* CNS leukemia allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT or AST no greater than 3 times ULN
* Chronic hepatitis allowed

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No active heart disease
* No myocardial infarction within the past 3 months
* No symptomatic coronary artery disease
* No arrhythmias uncontrolled by medication
* No uncontrolled congestive heart failure

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No persistent chronic toxic effects from prior chemotherapy greater than grade 1
* No uncontrolled active infection

  * Infections under control and under active treatment with antibiotics allowed

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 48 hours since prior hydroxyurea

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 2 weeks since prior myelosuppressive cytotoxic agents (in the absence of rapidly progressing disease)
* No other concurrent standard or investigational treatment for leukemia
* No concurrent disulfiram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Primary Completion 2004-09 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, MD, Study Chair — Vion Pharmaceuticals
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Giles F, Verstovsek S, Thomas D, Gerson S, Cortes J, Faderl S, Ferrajoli A, Ravandi F, Kornblau S, Garcia-Manero G, Jabbour E, O'Brien S, Karsten V, Cahill A, Yee K, Albitar M, Sznol M, Kantarjian H. Phase I study of cloretazine (VNP40101M), a novel sulfonylhydrazine alkylating agent, combined with cytarabine in patients with refractory leukemia. Clin Cancer Res. 2005 Nov 1;11(21):7817-24. doi: 10.1158/1078-0432.CCR-05-1070. PMID 16278404
- [Result] Giles FJ, Verstovsek S, Cortes J, et al.: Phase I study of VNP40101M (101M) and AraC in patients (pts) with refractory leukemia. [Abstract] J Clin Oncol 22 (14 Suppl): A-6617, 586s, 2004.